CLINICAL TRIAL: NCT06894212
Title: A Phase 3, Randomized, Double-blind, Parallel-group, Placebo-controlled, Multicenter Trial to Evaluate the Efficacy and Safety of SEP-363856 in Acutely Psychotic Participants With Schizophrenia
Brief Title: A Trial of the Efficacy and Safety of SEP-363856 in Acutely Psychotic Participants With Schizophrenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 382-201-00035
Record Dates: First submitted 2025-02-27; First posted 2025-03-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- SEP-363856 75 mg (Experimental): SEP-363856 75 mg/day
  Interventions: Drug: SEP-363856
- SEP-363856 100 mg (Experimental): SEP-363856 100 mg/day
  Interventions: Drug: SEP-363856

INTERVENTIONS:
Drug: SEP-363856 — tablet
  Arms: SEP-363856 100 mg; SEP-363856 75 mg
Other: Placebo — tablet
  Arms: Placebo

SUMMARY:
Evaluate the efficacy and safety of Ulotaront (SEP-363856) in acutely psychotic subjects with schizophrenia

DETAILED DESCRIPTION:
A Phase 3, Randomized, Double-blind, Parallel-group, Placebo-controlled, Multicenter Trial to Evaluate the Efficacy and Safety of SEP-363856 in Acutely Psychotic Participants with Schizophrenia

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female participants between 18 to 65 years of age (inclusive) at the time of consent.
* Participant has an identified reliable informant (eg, caregiver, relative, friend, case worker, residential treatment staff).
* Participant is experiencing an acute exacerbation or relapse of symptoms, with onset ≤ 2 months prior to screening

  1. The participant requires hospitalization for this acute exacerbation or relapse of symptoms.
  2. If already an inpatient at screening, has been hospitalized for less than 2 weeks for the current exacerbation at the time of screening.
* Participants who are experiencing an acute exacerbation of psychotic symptoms and marked deterioration of usual function as demonstrated by meeting ALL of the following criteria at the screening and baseline visits:

  1. Participant must have a PANSS total score ≥ 80

     AND
  2. Participant must have a CGI-S score ≥ 4.
* Participants who have received previous outpatient antipsychotic treatment at an adequate dose (minimal recommended dose for the treatment of schizophrenia according to the manufacturer labeling) for an adequate duration (at least 6 weeks) and who showed a previous good response.

Key Exclusion Criteria:

* Sexually active participants or persons of childbearing potential who do not agree to practice 2 different clinical trial sponsor approved methods of birth control or remain abstinent during the course of the trial and for 30 days after the last dose of study drug.
* Participant has a current DSM-5 diagnosis or presence of symptoms consistent with a DSM-5 diagnosis other than schizophrenia.
* Participant has had psychiatric hospitalization(s) for more than 30 days (cumulative) during the 90 days prior to screening.
* Participant has previously received SEP-363856 or was previously enrolled in a SEP-363856 clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in Positive And Negative Syndrome Scale (PANSS) total score at Week 6 | Baseline to Week 6
  To evaluate the efficacy of SEP-363856 (75 and 100 mg/day) compared with placebo in acutely psychotic participants with schizophrenia.
  PANSS total - 30-210 Higher score is indicative of greater symptomatology

SECONDARY OUTCOMES:
Clinical Global Impression-Severity (CGI-S) | Baseline to Week 6
  Change from baseline in CGI-S score at Week 6.
  CGI-S is 0-7 with higher score is indicative of greater symptomatology

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Pillar Clinical Research LLC - Bentonville Site # 145, Bentonville, Arkansas
  - Pillar Clinical Research (Little Rock AR) Site #153, Little Rock, Arkansas
  - Woodland International Research Group Site #141, Little Rock, Arkansas
  - Woodland Research Northwest Site # 138, Rogers, Arkansas
  - Clinical Innovations, Inc. dba CITrials (Bellflower) Site #131, Bellflower, California
  - ProScience Research Group Site #134, Culver City, California
  - CenExel CNS - Garden Grove (Collaborative Neuroscience Research) Site #123, Garden Grove, California
  - Synergy San Diego Site #128, Lemon Grove, California
  - Catalina Research Institute Site #142, Montclair, California
  - Clinical Innovations Inc. DBA CITrials (Riverside) Site #151, Riverside, California
  - Richmond Behavioral Associates LLC Site # 136, Riverside, California
  - CNRI - San Diego LLC Site # 126, San Diego, California
  - Schuster Medical Research Institute Site # 130, Sherman Oaks, California
  - CenExel CNS - Los Alamitos (Collaborative Neuroscience Research) Site #149, Torrance, California
  - Galiz Research Site #146, Hialeah, Florida
  - Segal Trials - Larkin Behavioral Health - Inpatient & Early Phase Site #147, Hollywood, Florida
  - Cenexel RCA (Research Centers of America) Site #124, Hollywood, Florida
  - Premier Clinical Research Institute - Site #150, Miami, Florida
  - D & H National Research Centers NC Site #143, Miami, Florida
  - Innovative Clinical Research, Inc. Site # 125, Miami Lakes, Florida
  - Health Synergy Clinical Research LLC Site #140, West Palm Beach, Florida
  - Synexus Clinical Research US Inc - Atlanta Site #148, Atlanta, Georgia
  - CenExel ACMR (Atlanta Center for Medical Research, LLC) Site #122, Atlanta, Georgia
  - CenExel IRA (CenExcel iResearch, LLC) Site #132, Decatur, Georgia
  - Accelerated Clinical Trials in Peachtree Corners GA Site # 127, Peachtree Corners, Georgia
  - Uptown Research Institute Site # 121, Chicago, Illinois
  - Pillar Clinical Research LLC (Chicago) Site #144, Chicago, Illinois
  - Eastern Clinical Research Associates - Site # 156, New Orleans, Louisiana
  - Cenexel CBH (CBH Health) Site # 129, Gaithersburg, Maryland
  - Hassman Research Institute, LLC Site #120, Marlton, New Jersey
  - Neuro-Behavioral Clinical Research Site # 135, Canton, Ohio
  - Community Clinical Research Inc Site # 133, Austin, Texas
  - InSite Clinical Research Site #152, DeSoto, Texas
  - HD Research - Memorial Hermann Surgery Center Memorial Village Site #137, Houston, Texas
  - Pillar Clinical Research LLC (Richardson, TX) Site #155, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the result of this study will be shared with researchers to achieve aims pre-specified in a methodology sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: http://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com